CLINICAL TRIAL: NCT04846764
Title: Rapid Declarative Neocortical Declarative Learning in Aging and Memory
Brief Title: Rapid Declarative Neocortical Declarative Learning in Aging and Memory Diseases (ANéRAVIMM)
Acronym: ANéRAVIMM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC20_9796_ANéRAVIMM
Record Dates: First submitted 2020-12-22; First posted 2021-04-15 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Neurological Diseases; Central Nervous System
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Active Comparator): 60 healthy volunteers (aged 18-40 and 60-80) will undergo an inclusion visit in order to check inclusion and non inclusion criteria.
  Then will be performed:
  Visit 1
  * Neuropsychological tests
  * A cranial MRI
  Visit 2
  • Neuropsychological tests
  Interventions: Other: Neuropsychological tests
- Patients with neurological diseases of the central nervous system (Experimental): 36 patients will undergo an inclusion visit in order to check inclusion and non inclusion criteria.
  Then will be performed:
  Visit 1
  * Neuropsychological tests
  * A cranial MRI
  Visit 2
  • Neuropsychological tests
  Interventions: Other: Neuropsychological tests

INTERVENTIONS:
Other: Neuropsychological tests — Scales and tests to evaluate:
  * laterality
  * anxiety
  * depression
  * professional level
  * education level
  * pre-morbid level
  * memory disorders
  Experimental procedure

SUMMARY:
Learning a person's name, new words, or simply remembering where the last conversation with a friend was held are examples of associative memory, frequently disturbed in brain pathologies, but also by aging. Although typically dependent on the hippocampus in the brain, a series of findings suggest that associative memory may persist, under certain circumstances, despite hippocampal damage. The ANéRAVIMM project aims to reveal this learning system, its cognitive and cerebral bases, and to evaluate its potential in patients with memory disorders.

DETAILED DESCRIPTION:
Three experimental cognitive tasks will be used in the ANéRAVIMM study. The first two tasks have been selected based on the literature and previous work of CHU Rennes team. They are two experiments that have produced promising results concerning the existence of a rapid neocortical learning system in declarative memory, and have in common the use of prior knowledge to promote learning.

In the first part of the study, these two tasks will be put in competition for their resistance to the effects of age. Brain aging is characterized by its deleterious impact on hippocampal functioning, and memory aging leads to an alteration of associative memory. Therefore, this first part will allow the learning paradigm that presents the best potential in brain-damaged patients to be retained in the second part of the ANéRAVIMM study.

The third task stems from recent work by CHU Rennes team in collaboration with Dr. Besson of the University of Liege, in the context of a very recent model of memory. It aims at estimating the ability to develop a representation of visual objects in memory at the entity level, i.e. an integrated representation, unifying all the perceptual, conceptual and contextual features of perceived information. This task has been adapted for the ANéRAVIMM project in order to test the hypothesis that this mnemonic representational level of the entity in memory could support rapid neocortical associative learning in declarative memory.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers

* aged 18 to 40 years old and aged 60 to 80 years old
* native French speaker
* right-handed
* with a level of education greater than or equal to the Certificate of Primary Education
* free of any medical or psychiatric condition that may interfere with cognition

Neurological patients

* patients with mild neurocognitive impairment due to Alzheimer's disease
* patients with semantic dementia syndrome
* right-handed patients with a right or left unilateral surgical lesion of the anterior temporal lobe as a result of pharmaco resistant temporal epilepsy, with no seizures in the last 6 months, with a memory quotient greater than 75, and free of internal extra temporal lesions on MRI
* patients with autoimmune limbic encephalitis who have been seizure-free for one month
* 1 KA patient, suffering from the rare syndrome of developmental amnesia

Exclusion Criteria:

All participants

* MRI contraindications
* sensory deficit interfering with experimental tests
* protected major (safeguard justice, trusteeship and guardianship) and persons deprived of liberty

Healthy volunteers

- deficit score on the MoCA scale according to current calibrations

Neurologic patients

* 7-items modified Hachinski ischemic score >2
* dementia
* epileptic seizure in the month prior to inclusion for epileptic patients undergoing surgery and limbic encephalitis patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-05-28 (Estimated); Study Completion 2024-05-28 (Estimated)

PRIMARY OUTCOMES:
Difference between young and old healthy subjects in experimental associative memory scores | Up to 1 month (time to perform the second visit)
Difference between healthy subjects and patients with SSHA damage in experimental associative memory scores | Up to 1 month (time to perform the second visit)
Correlations between SSHA volumes and experimental associative memory scores in healthy subjects and patients with SSHA damage | Up to 1 month (time to perform the second visit)
Correlations between rest-related functional connectivity within the Medial Temporal Lobes and experimental associative memory scores in healthy subjects | Up to 1 month (time to perform the second visit)

SECONDARY OUTCOMES:
Presence of significant correlations between memory scores for entity-level mnemonic representations and experimental associative memory scores in healthy subjects | Up to 1 month (time to perform the second visit)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France